CLINICAL TRIAL: NCT06121128
Title: The Effects of Inspiratory Muscle Training on Endurance Performance in Trained Athletes Under Normoxic and Hypoxic Conditions: A Gender-based Comprehensive Study
Acronym: RespiPerf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Gregoire Millet, Prof Ordinaire, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01638
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hypoxia, Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT): with a Female Control Group (FCON), a Male Control Group (MCON), a Female Training Group (FTRAIN), a Male Training Group (MTRAIN)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female Control Group (FCON) (Sham Comparator): female endurance trained athletes between 18 and 44 years old
  Interventions: Procedure: Normal Breathing
- Female Training Group (FTRAIN) (Experimental): female endurance trained athletes between 18 and 44 years old
  Interventions: Procedure: Inspiratory Muscle Training (IMT)
- Male Control Group (MCON) (Sham Comparator): male endurance trained athletes between 18 and 44 years old
  Interventions: Procedure: Normal Breathing
- Male Training Group (MTRAIN) (Experimental): male endurance trained athletes between 18 and 44 years old
  Interventions: Procedure: Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Procedure: Inspiratory Muscle Training (IMT) — The POWERbreathe™ Plus: an Inspiratory Muscle Training device (IMT) with adjustable resistance.
  Intervention lasts 4 weeks, with a frequency of 6 days/week, 2 series of 30 inspirations in the morning and evening.
  Resistance based on 60% of the Pressure Maximal Inspiratory (PMI). Progressive increase in resistance every week.
  Other Names: IMT
  Arms: Female Training Group (FTRAIN); Male Training Group (MTRAIN)
Procedure: Normal Breathing — No IMT performed
  Arms: Female Control Group (FCON); Male Control Group (MCON)

SUMMARY:
The POWERbreathe™ Plus: an Inspiratory Muscle Training device (IMT) with adjustable resistance.

Intervention lasts 4 weeks, with a frequency of 6 days/week, 2 series of 30 inspirations in the morning and evening.

Resistance based on 60% of the Pressure Maximal Inspiratory (PMI). Progressive increase in resistance every week.

Four laboratory visits: 2 pre-tests and 2 post-tests. Each pre- / post- test will go under normoxic and hypoxic conditions.

Measurements include Pulmonary functions (spirometry test); blood microcirculation (vascular occlusion test); gas exchanges (e.g. VO2max), cardiac parameters, heart rate variability, maximal aerobic power (incremental and time limit test)

DETAILED DESCRIPTION:
The POWERbreathe™ Plus: an Inspiratory Muscle Training device (IMT) with adjustable resistance.

Intervention lasts 4 weeks, with a frequency of 6 days/week, 2 series of 30 inspirations in the morning and evening.

Resistance based on 60% of the Pressure Maximal Inspiratory (PMI). Progressive increase in resistance every week.

Four laboratory visits: 2 pre-tests and 2 post-tests. Each pre- / post- test will go under normoxic and hypoxic conditions.

Measurements include Pulmonary functions (spirometry test); blood microcirculation (vascular occlusion test); gas exchanges (e.g. VO2max), cardiac parameters, heart rate variability, maximal aerobic power (incremental and time limit test)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion: endurance trained athletes between 18 and 44 years old

Exclusion Criteria:

cardiovascular, metabolic and respiratory diseases, smoking history, prescription medication (Two medication families are known to interfere with FC:

* Calcium channel blockers
* Beta-blockers

Two families are known to interfere during spirometry measurements:

* Inhaled beta-agonists
* Inhaled glucocorticoids)

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
sex-differences | One week prior and in the week immediately following the intervention
  Primary objective:
  To assess the change of a time limit duration in ergocycle after 4 weeks of inspiratory muscle training (IMT) between males and females.
Effect in hypoxia | One week prior and in the week immediately following the intervention
  Secondary objective:
  To assess the change of a time limit duration in ergocycle after 4 weeks of inspiratory muscle training (IMT) between hypoxia and normoxia.

IPD SHARING:
Plan to Share IPD: No